CLINICAL TRIAL: NCT05516368
Title: Psychological Monitoring of Victims of Terrorism and Effectiveness of Psychological Treatments.
Brief Title: TF-CBT for Long-term PTSD, Major Depressive Disorder and Anxiety Disorders in Victims of Terrorism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Spanish Association of Victims of Terrorism (Unknown)
Responsible Party: Principal Investigator, María de la Paz García Vera, Full-professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSI 2011-26450
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Posttraumatic Stress Disorder; Major Depressive Disorder; Anxiety Disorders
Keywords: Terrorism; Cognitive Behavior Therapy; Posttraumatic Stress Disorder (PTSD); Major Depression; Anxiety Disorders; Randomized Clinical Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TF-CBT (Experimental): 16 sessions of trauma-focused CBT adapted to victims of terrorism with long-term PTSD, major depressive disorder and/or anxiety disorders
  Interventions: Behavioral: TF-CBT
- Waiting list control (No Intervention): 4 months of waiting list condition

INTERVENTIONS:
Behavioral: TF-CBT — Modular TF-CBT therapy programme of 16 weekly individual sessions, each lasting 60-90 minutes.
  Arms: TF-CBT

SUMMARY:
The objective of this study is to test the efficacy of a Trauma-Focused Cognitive-Behavioural Therapy (TF-CBT) adapted for use with victims of terrorism in Spain who are diagnosed with posttraumatic stress disorder (PTSD), major depressive disorder and/or anxiety disorders subsequent to direct or indirect exposure to a series of terrorist attacks that occurred 20 years prior to treatment on average.

Spanish victims who meet the criteria for long-term posttraumatic stress disorder, major depressive disorder, and/or anxiety disorders related to direct or indirect exposure to terrorist attacks that occurred 20 years ago, on average, will be randomly assigned to 16 weekly sessions of TF-CBT (experimental group) or waiting list control (control group) conditions.

Between groups comparisons related to diagnostic rates and posttraumatic, depressive and anxiety symptoms will be made immediately after the intervention. Pre- follow-up comparisons related to diagnostic rates and posttraumatic, depressive, and anxiety symptoms will be carried out for the experimental group.

It is hypothesised that participants receiving TF-CBT will have significantly lower diagnostic rates and mean levels of posttraumatic, depressive and anxiety symptoms than the control group immediately after the intervention, and that they will experience significant pre-treatment to 6-month follow-up decreases in diagnostic rates and in posttraumatic, depressive and anxiety symptoms.

DETAILED DESCRIPTION:
This study will be a randomised, controlled, single-blind, single-center, and superiority trial, with two parallel groups (treatment and waiting list) and a primary endpoint based on the percentages of posttraumatic stress disorder, major depressive disorder and/or anxiety disorders, in the post-treatment (primary outcome). Mean levels of posttraumatic, depressive and anxiety symptoms in the post-treatment for both experimental and control groups, and changes in diagnostic percentages and in posttraumatic, depressive, and anxiety symptoms from baseline to 6-month follow-up for the experimental group are considered as secondary outcomes.

Researchers will contact the members of the Spanish Association of Victims of Terrorism and will invite them to an in-person diagnostic interview (pre-treatment evaluation) at a Spanish university. Eligible victims who meet the criteria for long-term posttraumatic stress disorder, major depressive disorder, and/or anxiety disorders will be randomly assigned to either experimental or control conditions. Random numbers generated by the Research Randomizer (Version 4.0) program (Urbaniack & Plous, 2013) will be used to assign subjects to treatment conditions. Randomisation will be performed as a block with a 1:1 allocation. As part of the informed consent process, the eligible individuals will be told that they will be enrolled in a free and voluntary psychological treatment programme, remaining blind to their allocation to the experimental or control group. Both groups will receive TF-CBT, although the experimental group will do it immediately and the control group, after 4 months of waiting list condition.

The modular TF-CBT therapy programme applied in this study will consist of 16 weekly individual sessions, each lasting 60-90 minutes. It will be organized around a structured protocol and the therapist will have a "checklist" of objectives to be fulfilled within each session. The core treatment component will be exposure, based on the application of Foa's "prolonged exposure" protocol (Foa et al., 2007), but adding specific techniques to control both depressive and anxiety disorders (i.e., progressive muscle relaxation, deep breathing exercises and pleasant activities scheduling), and cognitive restructuring all along the intervention. The TF-CBT intervention will be administered by a team of psychologists with a completed postgraduate training in clinical psychology and/or general health psychology, as well as a specific training in the provision of TF-CBT to victims of terrorism. The therapists will be supervised by senior clinical psychologists and will be monitored weekly.

Calculation of the sample size will be based on diagnostic percentages (dichotomous primary outcome), with a superiority margin of 5% between the two trial arms. In order to achieve an 80% power at the 5% level of significance with equal allocation, the total sample size should be N = 140 (n = 70 in each group). However, taking into account an average drop-out rate of 23.5% in the efficacy studies conducted on victims of terrorism (Garcia-Vera et al., 2015), the aim will be to recruit N = 184.

Contingency tables and chi2 tests will be used to assess post-treatment differences between the experimental vs. control groups in the percentage of individuals meeting diagnostic criteria for posttraumatic stress disorder, major depressive disorder and anxiety disorders, the primary endpoint. The McNemar's test will be carried out for two related samples to compare the percentage of those diagnosed in the pre-treatment and in the follow-up for the experimental group.

To compare the post-treatment symptomatology level of the two groups (treatment and control), analysis of variance will be carried out with repeated measurements on each of the symptomatology measures (posttraumatic, depressive and anxiety), in which the within-subject factor will be the time (pre-treatment and post-treatment), and the between-subject factor will be the experimental condition. As effect sizes, partial eta squared and Hedge's g between two groups at post-treatment will be calculated. Moreover, a pre-follow-up analyses of the symptomatology will be conducted for the experimental group and using repeated measures t-tests, and Hedge's g between pre and follow-up will be also calculated as effect sizes.

Following the approach of Jacobson & Truax (1991) to examine clinically significant changes, the percentages of patients in each group whose score in the post-treatment (or the follow-up) would be below the cut-off score that marked the step from clinically-significant symptomatology to "sub-syndromal" (the "C-score") will be calculated. This is 29 points for the Posttraumatic Stress Disorder Checklist, specific version (Sanz & García-Vera, 2015) and 14 for the Beck Depression Inventory-II and the Beck Anxiety Inventory. The Reliable Change Index will be also used (Jacobson & Truax, 1991; Mcglinchey et al., 2002). According to the Reliable Change Index data calculated by Sanz (2013, 2014; Sanz & García-Vera, 2015) for the Spanish population, the disorders of the patients whose scores drop by 12 points or more for the Posttraumatic Stress Disorder Checklist, specific version, or 10 points or more in the Beck Anxiety and Depression Inventories, will be designated as "improved". The chi2 tests will be carried out to examine differences between the experimental and control groups for each of these indices of clinical significance.

Per-protocol analyses will be conducted with the completers and Intention-to-treat analyses will be conducted considering all the participants initially enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being a direct victim of terrorism and/or a relative of someone killed or injured in a terrorist attack.
* Being of legal age
* Living in the same city or nearby
* Being diagnosed with PTSD, major depressive disorder, and/or anxiety disorders based on Diagnostic and Statistical Manual (DSM-IV) criteria (American Psychiatric Association, 2000).

Exclusion Criteria:

* Psychological condition unrelated to a terrorist attack
* Psychiatric emergency
* Declining to participate in the intervention before being diagnosed
* Medical contraindication(s) likely to interfere with treatment effectiveness, including organic brain syndrome, severe cognitive or sensor impairment, current substance use disorder, active psychotic or bipolar disorder, or severe dissociative amnesia
* Ongoing, in-process trauma-focused psychotherapy
* Inability to attend treatment sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of PTSD, depressive and anxiety disorders | Immediately after the intervention
  Percentage of PTSD, major depressive disorder and anxiety disorders, obtained by The Spanish version of the Structured Clinical Interview for DSM-IV, modules F and A (First et al., 1999).

SECONDARY OUTCOMES:
Post-traumatic stress symptoms | Immediately after the intervention
  Mean level of post-traumatic stress symptoms, measured by The Spanish version of the Posttraumatic Stress Disorder Checklist, specific version (PCL-S) (Vazquez et al.,2006).
Major depressive disorder symptoms | Immediately after the intervention
  Mean level of depressive symptoms, measured by the Spanish version of the Beck Depression Inventory-II (BDI-II) (Beck et al., 2011).
Anxiety symptoms | Immediately after the intervention
  Mean level of anxiety symptoms, measured by the Spanish version of the Beck Anxiety Inventory (BAI) (Beck & Steer 2011).
Change from Baseline Diagnosis of PTSD, depressive and anxiety disorders at 6 months | Baseline, 6 months
  Change in percentages of PTSD, depressive and anxiety disorders from Baseline to 6-month follow-up (obtained by The Spanish version of the Structured Clinical Interview for DSM-IV, modules F and A; First et al., 1999).
Change from Baseline mean level of post-traumatic stress symptoms at 6 months | Baseline, 6 months
  Change in the mean level of post-traumatic stress symptoms from Baseline to 6-month follow-up (measured by The Spanish version of the Posttraumatic Stress Disorder Checklist, specific version-PCL-S; Vazquez et al.,2006).
Change from Baseline mean level of depressive symptoms at 6 months | Baseline, 6 months
  Change in the mean level of depressive symptoms from Baseline to 6-month follow-up (measured by the Beck Depression Inventory-II- BDI-II; Beck et al., 2011).
Change from Baseline mean level of anxiety symptoms at 6 months | Baseline, 6 months
  Change in the mean level of anxiety symptoms from Baseline to 6-month follow-up (measured by Beck Anxiety Inventory-BAI; Beck & Steer, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: María Paz García Vera, Professor, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paz Garcia-Vera M, Sanz J, Gutierrez S. A Systematic Review of the Literature on Posttraumatic Stress Disorder in Victims of Terrorist Attacks. Psychol Rep. 2016 Aug;119(1):328-59. doi: 10.1177/0033294116658243. Epub 2016 Jul 7. PMID 27388691
- [Background] Garcia-Vera MP, Sanz J, Sanz-Garcia A. Ten Things Every Psychologist Should Know About Treating Psychological Disorders in Victims of Terrorism. Psicothema. 2021 May;33(2):177-187. doi: 10.7334/psicothema2021.33. PMID 33879289
- [Background] Moreno N, Sanz J, Garcia-Vera MP, Gesteira C, Gutierrez S, Zapardiel A, Cobos B, Marotta-Walters S. Effectiveness of trauma-focused cognitive behavioral therapy for terrorism victims with very long-term emotional disorders. Psicothema. 2019 Nov;31(4):400-406. doi: 10.7334/psicothema2018.165. PMID 31634084
- [Background] Garcia-Vera, M. P., Moreno, N., Sanz, J., Gutierrez, S., Gesteira, C., Zapardiel, A., & Marotta, S. (2015). Eficacia y utilidad clínica de los tratamientos para las víctimas adultas de atentados terroristas: una revisión sistemática. [Efficacy and clinical utility (effectiveness) of treatments for adult victims of terrorist attacks: A systematic review]. Psicología Conductual- Behavioral Psychology, 23, 215-244.
- [Result] Gesteira, C., Garcia-Vera, M.P., & Sanz, J. (2028). Porque el Tiempo no lo Cura Todo Eficacia de la Terapia Cognitivo-conductual Centrada en el Trauma para el Estrés postraumático a muy Largo Plazo en Víctimas de Terrorismo. [Because time does not heal all wounds: Efficacy of trauma-focused cognitive behavioral therapy for very long-term posttraumatic stress in victims of terrorism]. Clínica y Salud, 29(1), 9-13.

DOCUMENTS (1):
  • Informed Consent Form (2011-10-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT05516368/ICF_000.pdf